CLINICAL TRIAL: NCT02367131
Title: Post Marketing Surveillance in Japan on Drug Use of JARDIANCE® Tablets in Elderly Patients With Type 2 Diabetes Mellitus
Brief Title: Daily Use of JARDIANCE® Tablets in Japanese Elderly Patients With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245.98
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- JARDIANCE®
  Interventions: Drug: JARDIANCE®

INTERVENTIONS:
Drug: JARDIANCE® — JARDIANCE®
  Other Names: Empagliflozin

SUMMARY:
Study to investigate the safety and efficacy of daily use of JARDIANCE® Tablets in Japanese elderly patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion criteria:

Male and female elderly patients (age 65 and over) with type 2 diabetes mellitus who have never been treated with JARDIANCE® Tablets before the enrolment and start taking JARDIANCE® Tablets within 3 months after launch in Japan

Exclusion criteria:

None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients start taking JARDIANCE® Tablets within 3 months after launch will be included.
Sampling Method: Non-Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2015-02-24 (Actual); Primary Completion 2016-09-27 (Actual); Study Completion 2016-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- NISND Center, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Post-Marketing-Surveillance was a prospective study using a continuous investigation system. Patients with type 2 diabetes mellitus were included in the surveillance.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the study. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
Groups:
- JARDIANCE®: Elderly (age 65 and over) patients with type 2 diabetes mellitus who had never received JARDIANCE® Tablets were administered JARDIANCE® Tablets within 3 months after launch in Japan. Patients were administered orally with the starting at lower dosages (10 mg) of JARDIANCE®. In patients tolerating JARDIANCE, the dose was increased to 25 mg.
Period: Overall Study
Arm/Group | JARDIANCE®
Started (Registered) | 419
Treated | 417
Completed | 197
Not Completed | 222
Not completed — Adverse Event | 64
Not completed — No visit since the first visit | 3
Not completed — Request by patient | 53
Not completed — Improvement/remission | 2
Not completed — No change/progressive disease | 78
Not completed — Other than stated above | 20
Not completed — Not treated | 2

BASELINE CHARACTERISTICS:
Population: Safety Set : This analysis set included all elderly patients who had received treatment of JARDIANCE® Tablet at least one time except those who were found to have no observation after enrolment.
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 414
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.8 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170
  Male | 244

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Adverse Drug Reactions (ADRs)
Description: ADRs were defined as those adverse events for which the causal relationship was considered "Possibility high " or "Possibility low" or "Unknown" by the principal investigator, where:
  * Possibility high: There is a reasonable causal relationship between JARDIANCE® tablets administered and the adverse events (AE);
  * Possibility low: It is probably/possibly that there is a reasonable causal relationship between JARDIANCE® tablets administered and the AE;
  * Unknown: Cannot be judged because information is insufficient or contradictory. Percentages were rounded to two decimal places.
Time Frame: From first drug administration until 7 days after last drug adminstration, up to 52 weeks.
Population: Safety set: This analysis set included all elderly patients who had received treatment of JARDIANCE® Tablet at least one time except those who were found to have no observation after enrolment.
Measure: Number; unit: Percentage of participants
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 414
Percentage of participants | 20.53

2. Secondary Outcome: Change From Baseline in HbA1c (%) at the Last Observation During the Observation Period
Description: Change from baseline in HbA1c (%) at the last observation during the observation period is reported. Change from baseline was calculated as: HbA1c value at the last observation - HbA1c baseline value.
Time Frame: Baseline and last observation on treatment, up to week 52.
Population: Efficacy Set: This analysis set was a subset of the safety set, which included all patients in the "safety set" except those who had no available efficacy data for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of haemoglobin A1c
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 385
percentage of haemoglobin A1c | -0.36 (1.03)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at the Last Observation During the Observation Period
Description: Change from baseline in fasting plasma glucose (FPG) at the last observation during the observation period.
  Change from baseline was calculated as: FPG value at the last observation - FPG baseline value.
Time Frame: Baseline and last observation on treatment, up to week 52.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 240
milligram/deciliter (mg/dL) | -8.4 (45.6)

ADVERSE EVENTS:
Time Frame: From first drug administration until 7 days after last drug adminstration, up to 52 weeks
Description: Safety Set: This analysis set included all elderly patients who had received treatment of JARDIANCE® Tablet at least one time except those who were found to have no observation after enrolment.
Arm/Group | JARDIANCE®
All-Cause Mortality (participants affected / at risk) | 1/414
Serious Adverse Events (participants affected / at risk) | 6/414
Other Adverse Events (participants affected / at risk) | 0/414
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JARDIANCE® (N=414)
Atrial flutter (Cardiac disorders) | 1
Stress cardiomyopathy (Cardiac disorders) | 1
Age-related macular degeneration (Eye disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 1
Blood glucose increased (Investigations) | 1

LIMITATIONS AND CAVEATS:
The study was conducted in an unblinded manner and without controls. The sample size was not sufficient for rare ADRs. Some priority survey items were not reported, therefore incidence could not be estimated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No